CLINICAL TRIAL: NCT06443814
Title: A Clinical Trial on the Prevention of Coronary Artery Disease, Insulin Resistance and Hyperlipidemia in Black Women With Meditation and Health Education
Brief Title: Multicenter Trial of Meditation and Health Education for Cardiometabolic Disease in Black Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Schneider, MD (Other)
Collaborators: Morehouse School of Medicine (Other); Howard University (Other)
Responsible Party: Sponsor-Investigator, Robert Schneider, MD, Director, Institute for Natural Medicine and Prevention, Maharishi International University
Organization: Maharishi International University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1P50AT000082-03 (NIH)
Record Dates: First submitted 2023-11-13; First posted 2024-06-05 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Atherosclerotic Cardiovascular Disease; Metabolic Syndrome
Keywords: Meditation; Transcendental Meditation; Health Education; Prevention; Health Disparities; Women's Health
MeSH Terms: conditions — Atherosclerosis; Metabolic Syndrome; Health Education | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: This was a phase 2 randomized controlled trial of two behavioral interventions-Meditation and Health Education.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators, data collectors and usual medical providers were blinded to participant treatment status. Participants in both intervention groups were given similar expectations of positive outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcendental Meditation (Experimental): The TM technique is practiced for 20 minutes twice a day. Participants were instructed by a certified teacher in 7-step course to learn how to meditate according to previously standardized and validated procedures.
  Interventions: Behavioral: Transcendental Meditation
- Health Education (Active Comparator): The health education group was matched for instructor time and attention to the TM group. The classroom-based health education group received AHA-based guidelines for healthy diet, exercise and control of substance use. No stress management techniques are taught in this group.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Health Education — This was a didactic classroom-based control which educates the patient on adapting a healthier lifestyle through proper diet, exercise, and moderating substance usage according to current AHA guidelines. This intervention does not include a stress management component.
  Other Names: HE
  Arms: Health Education
Behavioral: Transcendental Meditation — TM was taught in a standardized and validated format as a simple, natural mental technique practiced for 20 minutes twice a day (morning and evening) to give rest and relaxation to mind and body. TM was taught by a certified instructor and a 7-step process taking place over 4 consecutive days after which the meditator can practice at home twice a day.
  Other Names: TM technique, TM
  Arms: Transcendental Meditation

SUMMARY:
This randomized controlled trial compared the efficacy of stress reduction with meditation to a health education (HE) group in 201 older African American women over a one-year study period. They were randomly allocated to either of two behavioral treatment groups-the Transcendental Meditation (TM) program or a health education (HE) program. Participants were recruited, tested, and instructed at two clinical sites: Howard University Hospital, Washington, DC and Morehouse (School of Medicine) Healthcare, Atlanta, GA. Main outcome measures were carotid intima-media thickness, insulin resistance, and behavioral factors.

DETAILED DESCRIPTION:
This was a randomized controlled trial that compared the effects of stress reduction using the Transcendental Meditation technique (TM) to a health education (HE) group in 201 African American women >55 years with CVD or at high CVD risk over a one-year intervention and follow-up period.

All participants were randomly allocated to either of two behavioral treatment groups-1) the Transcendental Meditation (TM) program or 2) a health education (HE) program of healthy diet, exercise and substance use control. Women participants were recruited, tested, and instructed at two sites:139 were recruited and randomized in Washington, DC and 61 in Atlanta, GA. Outcome measures were carotid intima-media thickness (IMT), insulin resistance, serum lipids, blood pressure and lifestyle (diet, exercise, substance use).

ELIGIBILITY:
Inclusion Criteria:

* African American women,
* 55 years or older with at least one of the five cardiovascular conditions (below):

Either/or:

* coronary heart disease or
* positive coronary angiography or
* previous MI or
* coronary revascularization or
* percutaneous transluminal coronary angioplasty (PTCA).

OR a risk factor assessment score of at least two points based on the Framingham study/ATP III report. Risk factors included diabetes, high systolic or diastolic BP, high cholesterol, high LDL-low HDL or smoking.

Exclusion Criteria:

Recent (last 3 months):

* myocardial infarction
* unstable angina
* coronary artery by-pass grafting (CABG)
* percutaneous transluminal coronary angioplasty (PTCA)
* stroke within the preceding three months
* carotid artery endarterectomy
* atrial fibrillation
* second or third degree AV block
* heart failure
* clinically significant valvular heart disease
* major psychiatric disorders,
* current alcohol/dependency disorder
* other drug abuse dependency disorder
* non-cardiac life-threatening illness
* participating in a formal stress management program
* plans to move out of the study area or travel extensively
* unwillingness to accept randomization into any study group.

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self identified women
Enrollment: 201 (Actual)
Dates: Start 2001-07 (Actual); Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Carotid intima-media thickness (CIMT) | 0 and 12 months
  B mode ultrasound measurement of carotid artery wall thickness

SECONDARY OUTCOMES:
Hemoglobin A1c | Before and after 12 months of intervention and follow up
  Hb1c as surrogate endpoint for diabetes
Insulin resistance | 0 and 12 months
  HOMA index utilizing glucose and insulin levels at timed intervals
Lipids | 0 and 12 months
  fasting levels of serum LDL, HDL, TC, TG
Blood pressure | 0, 4 and 12 months
  measured three times with a mercury sphygmomanometer 5 minutes apart and last two reading averaged
Physical Activity | 0, 4 and 12 months
  Exercise --using the Folsom Physical Activity Questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Linda Heaton, Study Director — Institute for Natural Medicine and Prevention, Maharishi International University
Locations (2):
- United States (2):
  - Howard University Heart Center, Washington D.C., District of Columbia
  - Morehouse School of Medicine - Morehouse Medical Associates, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No